CLINICAL TRIAL: NCT02657655
Title: Kinesia 360 Multi-Center Parkinson's Monitoring Study
Brief Title: Kinesia 360 Parkinson's Monitoring Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: University of South Carolina School of Medicine, Greenville (Unknown); University of Rochester (Other); Johns Hopkins University (Other); Prisma Health-Upstate (Other); National Institute on Aging (NIA) (NIH); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GLNT-K360-1; 5R44AG044293-04 (NIH); 5R44AG033947-05 (NIH); Pro000048239 (Other: IRB of the Greenville Health System)
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Dyskinesia; Tremor; Symptom Management; Technology; Wearable Sensors; Continuous Monitoring; Mobility
MeSH Terms: conditions — Parkinson Disease; Dyskinesias; Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Kinesia 360 Users (Experimental): Parkinson's patients will be monitored continuously using wearable Kinesia 360 sensors.
  Interventions: Device: Kinesia 360

INTERVENTIONS:
Device: Kinesia 360 — Kinesia 360 includes a mobile app and wireless motion sensors worn on the patient's wrist and ankle to quantify tremor, dyskinesias, and mobility throughout the day as he or she goes about normal activities. The app includes electronic diaries enable patients to rate their symptoms and log when medications are taken. Data is transferred to a cloud server where motor symptom reports are generated for clinician review.

SUMMARY:
Kinesia 360 is an ambulatory symptom monitoring device for Parkinson's Disease (PD). The aim of this study is to investigate the impact, validation, and usability of the Kinesia 360 system.

DETAILED DESCRIPTION:
This is a five-month study of 45 subjects (approximately 15 subjects per site), consisting of adult volunteers that have been clinically diagnosed with Parkinson's disease. Subjects will have a confirmed history of motor fluctuation with a variety of Parkinson's disease symptom severities. All subjects will user the Kinesia 360 system and complete motor diaries several times per month during the study period. Symptom reports will be provided to the treating clinical team. Motor function, quality of life, engagement, and satisfaction with care will be tracked throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease,
* History of motor fluctuations (2 hrs/day of Off time and/or 1 hr/day of troublesome dyskinesia)
* Fluent in English

Exclusion Criteria:

* Inability to carry out study activities
* Subjects with cognitive deficits that would prevent following instructions and serious medical conditions that would compromise a subject's safety
* Subjects who have dementia, exhibited by Montreal Cognitive Assessment (MoCa) score of 22 or less.
* Subjects who have had Deep Brain Stimulation (DBS) surgery less than 6 months prior to study enrollment, or who are deemed by the study investigator to be highly likely to undergo DBS surgery during the 6 month study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
% of assigned days with confirmed use | 5 months

SECONDARY OUTCOMES:
Diary measured Off time | 5 months
Diary measured On time with dyskinesia | 5 months
Off time as measured by Kinesia 360 | 5 months
On time with dyskinesia as measured by Kinesia 360 | 5 months
PDQ-39 responses | 5 months
Patient Assessment for Chronic Conditions (PACIC) responses | 5 months
Patient Activation Measure (PAM)-13 responses | 5 months
Number of clinic visits | 5 months
Number of patient/investigator communications | 5 months
Unified Parkinson's disease rating scale (UPDRS) | 5 months
Duration of time with patient | 5 months
Number and type of medication changes | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Heldman, PhD, Principal Investigator — Great Lakes NeuroTechnologies Inc.
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Rochester, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Greenville Health System, Greenville, South Carolina